CLINICAL TRIAL: NCT02651558
Title: Comparison of an Optical System to Continuously Measure Arterial Blood Pressure Against a Gold-standard Arterial Catheter
Brief Title: Optical System to Continuously Measure Arterial Blood Pressure
Acronym: BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BLOOD PRESSURE
Record Dates: First submitted 2015-12-17; First posted 2016-01-11 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OBPM 2015-MD-0022 - CHEST (Experimental): Cohort of 30 patients undergoing general anesthesia, monitored by optical signals at the chest
  Interventions: Device: Experimental: OBPM 2015-MD-0022 - CHEST
- OBPM 2015-MD-0022 - CHEST & FINGER (Experimental): Cohort of 10 patients undergoing general anesthesia, monitored by optical signals at the chest and at the fingertip
  Interventions: Device: Experimental: OBPM 2015-MD-0022 - CHEST & FINGER
- OBPM 2015-MD-0022 - FINGER (Experimental): Cohort of 30 patients undergoing general anesthesia, monitored by optical signals at the fingertip
  Interventions: Device: Experimental: OBPM 2015-MD-0022 - FINGER

INTERVENTIONS:
Device: Experimental: OBPM 2015-MD-0022 - CHEST — At the onset of general anesthesia:
  1. continuous measurements of radial arterial blood pressure values (arterial catheter, via a commercial PHILIPS IntelliVue MP50 monitor)
  2. continuous estimates of optical blood pressure values at the chest (optical blood pressure system, via Swissmedic approved OBPM measuring device 2015-MD-0022 developed by CSEM)
  will be recorded.
  Arms: OBPM 2015-MD-0022 - CHEST
Device: Experimental: OBPM 2015-MD-0022 - CHEST & FINGER — At the onset of general anesthesia:
  1. continuous measurements of radial arterial blood pressure values (arterial catheter, via a commercial PHILIPS IntelliVue MP50 monitor)
  2. continuous estimates of optical blood pressure values at the chest (optical blood pressure system, via Swissmedic approved OBPM measuring device 2015-MD-0022 developed by CSEM)
  3. continuous estimates of optical blood pressure values at the fingertip (optical blood pressure system, via Swissmedic approved OBPM measuring device 2015-MD-0022 developed by CSEM)
  will be recorded.
  Arms: OBPM 2015-MD-0022 - CHEST & FINGER
Device: Experimental: OBPM 2015-MD-0022 - FINGER — At the onset of general anesthesia:
  1. continuous measurements of radial arterial blood pressure values (arterial catheter, via a commercial PHILIPS IntelliVue MP50 monitor)
  2. continuous estimates of optical blood pressure values at the fingertip (optical blood pressure system, via Swissmedic approved OBPM measuring device 2015-MD-0022 developed by CSEM)
  will be recorded.
  Arms: OBPM 2015-MD-0022 - FINGER

SUMMARY:
Comparison of an optical method to continuously measure blood pressure against an invasive arterial catheter.

DETAILED DESCRIPTION:
The measurement of blood pressure during anesthesia is commonly performed by the inflation of a brachial cuff providing only intermittent blood pressure measurements. In some case, it is required to add a continuous invasive monitoring of blood pressure, via the insertion of an arterial catheter. Unfortunately, the related morbidity is not negligible. To limit the consequences of such a gesture, some developments have been done in the past to allow for continuous non-invasive measurements of blood pressure during anesthesia. Unfortunately, most of these devices are subject to important limitations and constraints of use.

A new system has been designed by CSEM consisting of an optical system fixed on patient's skin, absolutely non-invasive and easy to use. In order to study the reliability of this device, the investigators plan to compare its blood pressure estimates against gold-standard arterial catheter measurements during induction of general anesthesia on:

* 40 patients wearing the optical system at the chest.
* and 40 patients wearing the optical system at the fingertip

ELIGIBILITY:
Inclusion Criteria:

* patient requiring the placement of an arterial catheter for general anesthesia
* minimum of 18 years
* written consent

Exclusion Criteria:

* minor patient or incapable of discernment
* patient with AIMD
* thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Error (in mmHg) between paired determinations of arterial blood pressure from an optical device against reference measurements from an arterial catheter | 24 months
  The signals recorded by the optical blood pressure device will be retrospectively analysed (offline analysis) in order to test the hypothesis that blood pressure values as derived by the new device is comparable to blood pressure values as measured by an arterial catheter within the limits of agreement in mmHg stated by ISO 81060-2 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Ghamri Y, Proenca M, Hofmann G, Renevey P, Bonnier G, Braun F, Axis A, Lemay M, Schoettker P. Automated Pulse Oximeter Waveform Analysis to Track Changes in Blood Pressure During Anesthesia Induction: A Proof-of-Concept Study. Anesth Analg. 2020 May;130(5):1222-1233. doi: 10.1213/ANE.0000000000004678. PMID 32287129